CLINICAL TRIAL: NCT06397430
Title: Nutritional Support for Patients Operated on for Malignant Tumors of the Hepatico-pancreato-duodenal (HPD) Zone in the Early Postoperative Period
Brief Title: Nutritional Support for Patients Operated for Malignant Tumors in HPD Zone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaganda Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MUK_NutS-HPD-PO_2017
Record Dates: First submitted 2024-04-11; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Nutritional Support; Hepato-Biliary Neoplasm; Postoperative
Keywords: nutritional support; Hepato-Biliary Neoplasm; postoperative curation
MeSH Terms: interventions — Parenteral Nutrition; Enteral Nutrition

STUDY DESIGN:
Intervention Model Description: prospective, longitudinal, parallel study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - enteral nutrition (Experimental): patients receiving enteral nutrition (EN) after surgery
  Interventions: Dietary Supplement: enteral nutrition supplements
- Arm 2 - parenteral nutrition (Experimental): patients receiving parenteral nutrition (PN)
  Interventions: Dietary Supplement: parenteral nutrition supplements
- Arm 3 - mixed nutrition (Experimental): patients receiving mixed nutrition (MF)
  Interventions: Dietary Supplement: mixed nutrition supplements

INTERVENTIONS:
Dietary Supplement: parenteral nutrition supplements — parenteral nutrition
  Other Names: parenteral nutrition
  Arms: Arm 2 - parenteral nutrition
Dietary Supplement: enteral nutrition supplements — enteral nutrition
  Other Names: enteral nutrition
  Arms: Arm 1 - enteral nutrition
Dietary Supplement: mixed nutrition supplements — mixed nutrition
  Other Names: mixed nutrition
  Arms: Arm 3 - mixed nutrition

SUMMARY:
A comprehensive comparative analysis of the effectiveness of isolated enteral, isolated parenteral and mixed type of nutritional support in the early postoperative period in patients after operations performed on the malignant neoplasms of hepatico-pancreatico-duodenal zone.

DETAILED DESCRIPTION:
A prospective, longitudinal, parallel study and retrospective analysis of the results of treatment of 91 patients with malignant tumors of the hepatico-pancreato-duodenal zone who underwent the following operations:

1. resection of various segments of the liver;
2. hemihepatectomy;
3. transhepatic drainage of the right and left hepatic duct;
4. bypass gastroenteroanastomosis or cholecystenteroanastomosis with interintestinal enteroenteroanastomosis according to Brown;
5. gastro-pancreato-duodenal resection;
6. corpore-caudal resection of the pancreas with splenectomy.

The first group (n=31) included patients who received enteral nutrition (EN) after surgery. The second group (n=30) included patients who received parenteral nutrition (PN) and the third group (n=30) who received mixed nutrition (MN), as a variation of the partial parenteral nutrition technique, in the early postoperative period.

Some nutritional status indicators available for determination at the Oncology Clinic were assessed - body mass index (weight measurements were carried out before surgery, on the 5th, 10th and 15th days), basal metabolic rate (calculated using the Harris-Benedict equation, based on anthropometric data of the patient (gender, age, weight and height).), laboratory parameters: blood hemoglobin, lymphocytes, total protein, serum albumin, serum transferrin, total bilirubin and direct, alanine aminotransferase (ALT), aspartate aminotransferase (AST), which are related to the traditional method for assessing nutritional status

ELIGIBILITY:
Inclusion Criteria:

female and male patients in age of 20-75 with malignant tumors of the hepato-pancreato-duodenal zone who have undergone any of the following operations:

1. resection of various segments of the liver;
2. hemihepatectomy;
3. transhepatic drainage of the right and left hepatic duct;
4. bypass gastroenteroanastomosis or cholecystoenteroanastomosis with interintestinal enteroenteroanastomosis according to Brown;
5. gastro-pancreatoduodenal resection;
6. corporecaudal resection of the pancreas with splenectomy.

Exclusion Criteria:

* patients in age of up to 20 and older than 75
* pregnant and breastfeeding women

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants with changes of BMI in kg/m^2 | Day 0, Day 5, Day 10, Day15
  Variables of Body mass index measured by Canadian Guidelines for Body Weight Classification in Adults
Basal Metabolic rate | Day 0, Day 5, Day 10, Day15
  basal metabolic rate according to the Harris-Benedict equation
Total protein level in Blood | Day 0, Day 5, Day 10, Day15
  Blood biochemical analysis: total protein in g/L
Serum albumin in g/L | Day 0, Day 5, Day 10, Day15
  Blood biochemical analysis: serum albumin in g/L
Serum transferrin in g/L | Day 0, Day 5, Day 10, Day15
  Blood biochemical analysis: serum transferrin in g/L
Total bilirubin in mmol/L | Day 0, Day 5, Day 10, Day15
  Blood biochemical analysis: total bilirubin in mmol/L
Direct bilirubin in mmol/L | Day 0, Day 5, Day 10, Day15
  Blood biochemical analysis: direct bilirubin in mmol/L
ALT in IU/L | Day 0, Day 5, Day 10, Day15
  Blood biochemical analysis: ALT in IU/L
AST in IU/L | Day 0, Day 5, Day 10, Day15
  Blood biochemical analysis: AST in IU/L

CONTACTS AND LOCATIONS:
Overall Officials: Sherzad Davanov, MD, Principal Investigator — Karaganda Medical University
Locations (1):
- Karaganda Medical University, Karaganda, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT06397430/Prot_SAP_ICF_000.pdf